CLINICAL TRIAL: NCT02930018
Title: A Multicentre, Randomized, Double-blinded, Placebo-controlled, Parallel Group, Single-dose Design to Determine the Efficacy and Safety of Intravenous NA-1 in Subjects With Acute Ischemic Stroke Undergoing Endovascular Thrombectomy
Brief Title: Safety and Efficacy of Nerinetide (NA-1) in Subjects Undergoing Endovascular Thrombectomy for Stroke
Acronym: ESCAPE-NA1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NoNO Inc. (Industry)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA-1-007
Record Dates: First submitted 2016-10-06; First posted 2016-10-11 (Estimated); Results first posted 2020-12-14 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Stroke, Acute
Keywords: Acute Ischemic Stroke; Endovascular Thrombectomy; Neuroprotection; Tat-NR2B9c; NA-1; Nerinetide
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Drug vehicle only
  Interventions: Drug: Placebo
- Nerinetide (NA-1), 2.6 mg/kg (Experimental)
  Interventions: Drug: Nerinetide (NA-1), 2.6 mg/kg

INTERVENTIONS:
Drug: Nerinetide (NA-1), 2.6 mg/kg — Single intravenous infusion of nerinetide over 10 ± 1 minutes
  Other Names: NA-1
  Arms: Nerinetide (NA-1), 2.6 mg/kg
Drug: Placebo — Placebo Comparator: Placebo
  Other Names: Drug vehicle only
  Arms: Placebo

SUMMARY:
The ESCAPE-NA-1 study is designed to determine the safety and efficacy of the neuroprotectant, Nerinetide (NA-1), in reducing global disability in subjects with major acute ischemic stroke (AIS) with a small established infarct core and with good collateral circulation who are selected for endovascular revascularization.

DETAILED DESCRIPTION:
Trial Objectives:

The primary objective is to determine the efficacy of the neuroprotectant, Nerinetide, in reducing global disability in subjects with major acute ischemic stroke (AIS) with a small established infarct core and with good collateral circulation selected for rapid endovascular revascularization.

The secondary objectives are to determine the efficacy of Nerinetide in:

* Reducing functional dependence
* Improving neurological outcome
* Improving activities of daily living
* Reducing mortality rate The leading safety objectives are to determine the effect of administering a dose of 2.6 mg/kg (up to a maximum dose of 270 mg) intravenous (IV) infusion of Nerinetide to subject with acute stroke who are selected for endovascular revascularization on serious adverse events (SAEs) and 90-day mortality.

Trial Design:

This study is a Phase 3, randomized, multicentre, blinded, placebo-controlled, parallel group, single-dose design. Subjects harboring an acute ischemic stroke and who are selected for endovascular revascularization in accordance with local institutional practices and who harbor a small established infarct core and with good collateral circulation will be given a single, 2.6 mg/kg (up to a maximum dose of 270 mg) intravenous dose of Nerinetide (NA-1) or placebo as soon as they are deemed to have met the enrollment criteria and with the intention of starting administration within 30 minutes of randomization. The randomization will be by stochastic minimization to balance baseline factors.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke (AIS) for immediate endovascular treatment
2. Age 18 or greater.
3. Onset (last-seen-well) time to randomization time within 12 hours.
4. Disabling stroke defined as a baseline National Institutes of Health Stroke Score (NIHSS) > 5 at the time of randomization.
5. Pre-stroke (24 hours prior to stroke onset) independent functional status in activities of daily living with modified Barthel Index (BI) > 90 (95 or 100). Patient must be living in their own home, apartment or seniors lodge where no nursing care is required.
6. Confirmed symptomatic intracranial occlusion, based on multiphase or dynamic computerized tomographic angiography (CTA), at one or more of the following locations: Intracranial carotid T/L, M1 middle cerebral artery (MCA). Functionally, when defining the M1 or the M2, the bulk of the MCA territory must be ischemic.
7. Non-contrast computed tomography (NCCT) and CTA (multiphase or dynamic) for trial eligibility performed or repeated at ESCAPE-NA1 stroke centre with endovascular suite on-site.
8. Endovascular treatment with declared first endovascular approach as either stent retriever or aspiration device, and intended to be initiated (arterial access) within 60 minutes of baseline/qualifying NCCT and to first recanalization of 90 minutes. Study drug intended to be administered within 60 minutes of the baseline/qualifying NCCT.
9. Signed informed consent from subject or legally authorized representative or, if required to enable inclusion by applicable national laws and regulations and the applicable independent review boards/Ethics Committee requirements for obtaining consent, from the investigator after consultation with an independent physician who is not otherwise participating in the trial.

Exclusion Criteria:

1. Evidence of a large core of established infarction defined as ASPECTS 0-4.
2. Evidence of absence of collateral circulation on CTA (Collateral score of 0 or 1).
3. Intent to use any endovascular device other than a stent retriever or clot aspiration device or intra-arterial medications as the initial thrombectomy approach.
4. Intent to use any intravenous thrombolytic other than alteplase if intravenous thrombolysis is planned.
5. No femoral pulses, very difficult endovascular access or extreme tortuosity of great vessels that is predicted to result in an inability to deliver timely endovascular therapy. Direct common carotid or radial/brachial/axillary access is permissible.
6. Estimated or known weight > 120 kg or < 45 kg.
7. Pregnancy; if a woman is of childbearing potential a urine or serum beta human chorionic gonadotropin (β-hCG) test is positive, or breastfeeding.
8. Severe contrast allergy or absolute contraindication to iodinated contrast preventing endovascular intervention, including any contraindications listed in the prescribing information approved by local authorities (e.g., patients with decompensated heart failure as a contraindication for the use of VISIPAQUE™ 270 in Germany).
9. Clinical history, past imaging or clinical judgment suggests that the intracranial occlusion is chronic or there is suspected intracranial dissection such that there is a predicted lack of success with endovascular intervention.
10. Prior enrolment in the ESCAPE-NA1 trial or prior receipt of NA-1 for any reason.
11. Severe known renal impairment defined as requiring dialysis (hemo- or peritoneal) or if known a creatinine clearance < 29 mL/min.
12. Patient has a severe or fatal comorbid illness that will prevent improvement or follow-up.
13. Patient cannot complete follow-up treatment due to co-morbid non-fatal illness or they are known to be a visitor to the city or any other known reason for which follow-up would be impossible (e.g. incarcerated in a federal prison).
14. Participation in another clinical trial investigating a drug, medical device, or a medical procedure in the 30 days preceding study inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1105 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Hill, MD MSc, Principal Investigator — University of Calgary
Locations (50):
- United States (20):
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - California Pacific Medical Center - Davies Campus, San Francisco, California
  - Providence Little Company of Mary Medical Center Torrance, Torrance, California
  - Swedish Medical Center, Englewood, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Baptist Health Medical Center, Jacksonville, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - WellStar Health Systems, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - NYU Lutheran Medical Center, Brooklyn, New York
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Riverside Radiology, Columbus, Ohio
  - Abington Memorial Hospital, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Chattanooga Center for Neurologic Research, Chattanooga, Tennessee
  - Valley Baptist Medical Center, Harlingen, Texas
  - Swedish Medical Center- Cherry Hill Campus, Seattle, Washington
- Australia (2):
  - Royal Adelaide Hospital, Adelaide
  - Royal Melbourne Hospital, Parkville
- Canada (14):
  - University of Calgary - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver Stroke Program Research Office/ Vancouver General Hosptial, Vancouver, British Columbia
  - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre- University Hospital, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Centre, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario
  - CHUM Hopital Notre-Dame, Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - CHU de Quebec- Universite Laval- Hopital de l'Enfant-Jesus, Québec, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Germany (5):
  - Universitätsklinikum Carl Gustav Carus Dresdner Neurovaskulares Centrum, Dresden
  - Klinik für Radiologie und Neuroradiologie, Essen
  - University Medical Center Goettingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Neurologische Klinik, Universität Heidelberg, Heidelberg
- Ireland (2):
  - Beaumont Hospital, Dublin
  - Mater Hospital, Dublin
- South Korea (4):
  - Dongsan Medical Centre, Daegu
  - Inha University Hospital, Incheon
  - Samsung Medical Center, Seoul
  - Yonsei Univ, Severence, Seoul
- Sweden (2):
  - Skåne University Hospital, Lund
  - Karolinksa Institutet, Stockholm
- Royal Victoria Hospital, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hill MD, Martin RH, Mikulis D, Wong JH, Silver FL, Terbrugge KG, Milot G, Clark WM, Macdonald RL, Kelly ME, Boulton M, Fleetwood I, McDougall C, Gunnarsson T, Chow M, Lum C, Dodd R, Poublanc J, Krings T, Demchuk AM, Goyal M, Anderson R, Bishop J, Garman D, Tymianski M; ENACT trial investigators. Safety and efficacy of NA-1 in patients with iatrogenic stroke after endovascular aneurysm repair (ENACT): a phase 2, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2012 Nov;11(11):942-50. doi: 10.1016/S1474-4422(12)70225-9. Epub 2012 Oct 8. PMID 23051991
- [Background] Cook DJ, Teves L, Tymianski M. Treatment of stroke with a PSD-95 inhibitor in the gyrencephalic primate brain. Nature. 2012 Feb 29;483(7388):213-7. doi: 10.1038/nature10841. PMID 22388811
- [Background] Cook DJ, Teves L, Tymianski M. A translational paradigm for the preclinical evaluation of the stroke neuroprotectant Tat-NR2B9c in gyrencephalic nonhuman primates. Sci Transl Med. 2012 Oct 3;4(154):154ra133. doi: 10.1126/scitranslmed.3003824. PMID 23035045
- [Background] Sun HS, Doucette TA, Liu Y, Fang Y, Teves L, Aarts M, Ryan CL, Bernard PB, Lau A, Forder JP, Salter MW, Wang YT, Tasker RA, Tymianski M. Effectiveness of PSD95 inhibitors in permanent and transient focal ischemia in the rat. Stroke. 2008 Sep;39(9):2544-53. doi: 10.1161/STROKEAHA.107.506048. Epub 2008 Jul 10. PMID 18617669
- [Background] Aarts M, Liu Y, Liu L, Besshoh S, Arundine M, Gurd JW, Wang YT, Salter MW, Tymianski M. Treatment of ischemic brain damage by perturbing NMDA receptor- PSD-95 protein interactions. Science. 2002 Oct 25;298(5594):846-50. doi: 10.1126/science.1072873. PMID 12399596
- [Background] Sattler R, Xiong Z, Lu WY, Hafner M, MacDonald JF, Tymianski M. Specific coupling of NMDA receptor activation to nitric oxide neurotoxicity by PSD-95 protein. Science. 1999 Jun 11;284(5421):1845-8. doi: 10.1126/science.284.5421.1845. PMID 10364559
- [Background] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Result] Hill MD, Goyal M, Menon BK, Nogueira RG, McTaggart RA, Demchuk AM, Poppe AY, Buck BH, Field TS, Dowlatshahi D, van Adel BA, Swartz RH, Shah RA, Sauvageau E, Zerna C, Ospel JM, Joshi M, Almekhlafi MA, Ryckborst KJ, Lowerison MW, Heard K, Garman D, Haussen D, Cutting SM, Coutts SB, Roy D, Rempel JL, Rohr AC, Iancu D, Sahlas DJ, Yu AYX, Devlin TG, Hanel RA, Puetz V, Silver FL, Campbell BCV, Chapot R, Teitelbaum J, Mandzia JL, Kleinig TJ, Turkel-Parrella D, Heck D, Kelly ME, Bharatha A, Bang OY, Jadhav A, Gupta R, Frei DF, Tarpley JW, McDougall CG, Holmin S, Rha JH, Puri AS, Camden MC, Thomalla G, Choe H, Phillips SJ, Schindler JL, Thornton J, Nagel S, Heo JH, Sohn SI, Psychogios MN, Budzik RF, Starkman S, Martin CO, Burns PA, Murphy S, Lopez GA, English J, Tymianski M; ESCAPE-NA1 Investigators. Efficacy and safety of nerinetide for the treatment of acute ischaemic stroke (ESCAPE-NA1): a multicentre, double-blind, randomised controlled trial. Lancet. 2020 Mar 14;395(10227):878-887. doi: 10.1016/S0140-6736(20)30258-0. Epub 2020 Feb 20. PMID 32087818
- [Derived] Stebner A, Bosshart SL, Fujiwara S, Frei D, Tarpley J, Dowlatshahi D, Rempel JL, Hill MD, Goyal M, Ospel JM; ESCAPE-NA1 Investigators. Association of baseline infarct size, reperfusion grade and intracranial hemorrhage in patients undergoing thrombectomy. J Neurointerv Surg. 2025 Mar 23:jnis-2025-023103. doi: 10.1136/jnis-2025-023103. Online ahead of print. PMID 40122606
- [Derived] Ospel JM, Goyal M, Menon BK, Almekhlafi MA, Zerna C, Nogueira RG, McTaggart RA, Demchuk AM, Poppe AY, Rempel JL, Joshi M, Kashani N, Heard K, Field TS, Dowlatshahi D, van Adel B, Swartz RH, Shah R, Sauvageau E, Puetz V, Silver FL, Campbell B, Chapot R, Tymianski M, Hill MD; ESCAPE-NA1 Investigators. Factors Influencing Nerinetide Effect on Infarct Volume in Patients Without Alteplase in the Randomized ESCAPE-NA1 Trial. Stroke. 2025 Jan;56(1):14-21. doi: 10.1161/STROKEAHA.124.048601. Epub 2024 Dec 9. PMID 39648909
- [Derived] Ospel JM, Rex N, Rinkel L, Kashani N, Buck B, Rempel J, Sahlas D, Kelly ME, Budzik R, Tymianski M, Hill MD, Goyal M; ESCAPE-NA1 Investigators. Prevalence of "Ghost Infarct Core" after Endovascular Thrombectomy. AJNR Am J Neuroradiol. 2024 Mar 7;45(3):291-295. doi: 10.3174/ajnr.A8113. PMID 38272571
- [Derived] Fladt J, Guo J, Specht JL, Wang M, Chan LL, Mctaggart R, Buck BH, Aviv R, Swartz RH, Field TS, Tarpley J, Shah R, Goyal M, Tymianski M, Hill MD, Demchuk A, d'Esterre C, Barber P. Infarct Evolution on MR-DWI After Thrombectomy in Acute Stroke Patients Randomized to Nerinetide or Placebo: The REPERFUSE-NA1 Study. Neurology. 2024 Jan 23;102(2):e207976. doi: 10.1212/WNL.0000000000207976. Epub 2023 Dec 22. PMID 38165335
- [Derived] Singh N, Cimflova P, Ospel JM, Kashani N, Marko M, Mayank A, Hill MD; ESCAPE-NA1 Trial Investigators. Prevalence and Predictors of Multivessel Occlusions at Baseline Imaging in ESCAPE-NA1 Trial. Stroke. 2023 Jun;54(6):e233-e234. doi: 10.1161/STROKEAHA.123.043027. Epub 2023 May 11. No abstract available. PMID 37165867
- [Derived] Singh N, Cimflova P, Ospel JM, Kashani N, Marko M, Mayank A, Nogueira RG, McTaggart RA, Demchuk AM, Poppe AY, Rempel JL, Field TS, Dowlatshahi D, van Adel B, Swartz RH, Shah R, Sauvageau E, Puetz V, Silver FL, Campbell B, Chapot R, Tymianski M, Goyal M, Almekhlafi MA, Hill MD; ESCAPE-NA1 Trial Investigators. Infarcts in a New Territory: Insights From the ESCAPE-NA1 Trial. Stroke. 2023 Jun;54(6):1477-1483. doi: 10.1161/STROKEAHA.122.042200. Epub 2023 Apr 21. PMID 37082967

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with acute ischaemic stroke who were selected to undergo EVT (endovascular thrombectomy) were enrolled. The trial was done at acute care hospitals. Patients were randomly assigned (1:1) to receive a single intravenous dose of nerinetide (NA-1) or placebo. All patients underwent endovascular thrombectomy and received alteplase in usual care when indicated.
Pre-assignment Details: The trial drug was administered as soon as possible after randomisation.
Period: Overall Study
Arm/Group | Placebo | Nerinetide (NA-1), 2.6 mg/kg
Started | 556 | 549
Completed | 550 | 546
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nerinetide (NA-1), 2.6 mg/kg | Total
Number analyzed (Participants) | 556 | 549 | 1105
Age, Continuous [Median (Full Range); unit: years] | 70.0 [20 to 103] | 71.0 [18 to 98] | 70.0 [18 to 103]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 281 | 268 | 549
  Male | 275 | 281 | 556
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 8 | 23
  Not Hispanic or Latino | 540 | 541 | 1081
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Under 'Unknown or Not reported' category the number of participants for the 'Other' category is indicated
  Participants
    American Indian or Alaska Native | 2 | 2 | 4
    Asian | 52 | 55 | 107
    Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
    Black or African American | 31 | 45 | 76
    White | 453 | 436 | 889
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 15 | 11 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 252 | 253 | 505
  South Korea | 20 | 22 | 42
  Sweden | 8 | 6 | 14
  United States | 203 | 211 | 414
  Ireland | 5 | 4 | 9
  United Kingdom | 1 | 1 | 2
  Australia | 25 | 18 | 43
  Germany | 42 | 34 | 76
Alteplase Treatment [Count of Participants; unit: Participants] — Treatment with alteplase as part of standard-of-care in addition to study drug
  Participants
    Participants treated with alteplase | 329 | 330 | 659
    Participants not treated with alteplase | 227 | 219 | 446

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With mRS Score of 0 to 2
Description: Overall number of subjects experiencing a favorable functional outcome 90 days post-randomization, defined as 0 to 2 on the mRS.
  The modified Rankin Scale (mRS) is a valid and reliable clinician-reported measure of global disability that has been widely applied for evaluating recovery from stroke. It is a scale used to measure functional recovery (the degree of disability or dependence in daily activities) of people who have suffered a stroke. mRS scores range from 0 (best outcome) to 6 (worst outcome), with 0 indicating no residual symptoms; 5 indicating bedbound, requiring constant care; and 6 indicating death.
Time Frame: 90 Days
Population: Intent-to-Treat Population
Measure: Count of Participants; unit: Participants
Groups:
- Nerinetide, 2.6 mg/kg: Single intravenous infusion of nerinetide over 10 ± 1 minutes
Arm/Group | Placebo | Nerinetide, 2.6 mg/kg
Number analyzed (Participants) | 556 | 549
Participants | 329 | 337
Statistical Analysis 1: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; The primary hypothesis was that administration of nerinetide (NA-1) would result in an increase in the proportion of responders. The primary analysis was a Wald test for treatment group difference in the primary outcome from a logistic regression adjusted for the 2 stratification variables (alteplase use, first declared thrombectomy device), and the 6 covariates used in the minimization. The trial was designed to have 80% power to detect an 8.7% absolute difference between groups; Test type: Superiority — It is hypothesized that the cleavage of nerinetide by plasmin which is activated by tissue plasminogen activators, such as alteplase results in a treatment modification of nerinetide in AIS (Acute Ischemic Stroke) patients with prior administration of alteplase as part of standard-of-care; p = 0.335, Regression, Logistic — 2 sided 0.05 significance level; Odds Ratio (OR) = 1.146, 95% CI 2-sided [0.869 to 1.511]

2. Secondary Outcome: Number of Subjects With NIHSS Score of 0 to 2
Description: Number of subjects with good neurological outcome, as defined by a score of 0 to 2 on the NIHSS at Day 90 or the last rating.
  The National Institutes of Health Stroke Scale (NIHSS) is a standardized neurological examination score that is a valid and reliable measure of disability and recovery after acute stroke. Scores range from 0 to 42, with higher scores indicating increasing severity.
Time Frame: 90 Days or the last rating
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerinetide, 2.6 mg/kg
Number analyzed (Participants) | 556 | 549
Participants | 320 | 320
Statistical Analysis 1: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; Test type: Superiority — It is hypothesized that the cleavage of nerinetide by plasmin which is activated by tissue plasminogen activators, such as alteplase results in a treatment modification of nerinetide in AIS patients with prior administration of alteplase as part of standard-of-care; p = 0.866, Regression, Logistic — 2 sided 0.05 significance level; Odds Ratio (OR) = 1.024, 95% CI 2-sided [0.781 to 1.342]

3. Secondary Outcome: Mortality Rate
Description: Mortality rate, as defined by event rate (%) for mortality over the 90-day study period
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerinetide, 2.6 mg/kg
Number analyzed (Participants) | 556 | 549
Participants | 74 | 64
Statistical Analysis 1: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.199, Regression, Logistic — 2 sided 0.05 significance level; Odds Ratio (OR) = 0.776, 95% CI 2-sided [0.527 to 1.143]

4. Post Hoc Outcome: Number of Subjects With mRS Score of 0 to 2 in the No-alteplase Sub-group
Description: Overall number of subjects experiencing a favorable functional outcome 90 days post-randomization, defined as 0 to 2 on the mRS in the sub-group of participants not treated with alteplase as part of standard-of-care.
  The modified Rankin Scale (mRS) is a valid and reliable clinician-reported measure of global disability that has been widely applied for evaluating recovery from stroke. It is a scale used to measure functional recovery (the degree of disability or dependence in daily activities) of people who have suffered a stroke. mRS scores range from 0 (best outcome) to 6 (worst outcome), with 0 indicating no residual symptoms; 5 indicating bedbound, requiring constant care; and 6 indicating death.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerinetide, 2.6 mg/kg
Number analyzed (Participants) | 227 | 219
Participants | 113 | 130
Statistical Analysis 1: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; Test type: Superiority; p = 0.028, Regression, Logistic; Odds Ratio (OR) = 1.657, 95% CI 2-sided [1.055 to 2.603]
Statistical Analysis 2: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; Test type: Superiority; Absolute Risk Difference (%) = 9.6 — The unadjusted absolute risk difference in % between nerinetide and placebo in the no-alteplase subgroup
Statistical Analysis 3: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; Test type: Superiority; Relative Risk Difference (%) = 19.3 — The unadjusted relative risk difference in % between nerinetide and placebo in the no-alteplase subgroup

5. Post Hoc Outcome: Number of Subjects With NIHSS Score of 0 to 2 in the No-Alteplase Sub-group
Description: Number of subjects with good neurological outcome, as defined by a score of 0 to 2 on the NIHSS at Day 90 or the last rating in the sub-group of participants not treated with alteplase as part of standard-of-care.
  The National Institutes of Health Stroke Scale (NIHSS) is a standardized neurological examination score that is a valid and reliable measure of disability and recovery after acute stroke. Scores range from 0 to 42, with higher scores indicating increasing severity.
Time Frame: 90 days or last rating
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerinetide, 2.6 mg/kg
Number analyzed (Participants) | 227 | 219
Participants | 113 | 129
Statistical Analysis 1: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; Test type: Superiority; p = 0.088, Regression, Logistic; Odds Ratio (OR) = 1.482, 95% CI 2-sided [0.943 to 2.329]
Statistical Analysis 2: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; Test type: Superiority; Absolute Risk Difference (%) = 9.1 — The unadjusted absolute risk difference in % between nerinetide and placebo in the no-alteplase subgroup
Statistical Analysis 3: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; Test type: Superiority; Relative Risk Difference (%) = 18.3 — The unadjusted relative risk difference in % between nerinetide and placebo in the no-alteplase subgroup

6. Post Hoc Outcome: Mortality Rate in the No-Alteplase Sub-group
Description: Mortality rate, as defined by event rate (%) for mortality over the 90-day study period in the sub-group of participants not treated with alteplase as part of standard-of-care
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerinetide, 2.6 mg/kg
Number analyzed (Participants) | 227 | 219
Participants | 43 | 25
Statistical Analysis 1: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; Test type: Superiority; p = 0.055, Regression, Logistic; Odds Ratio (OR) = 0.572, 95% CI 2-sided [0.323 to 1.013]
Statistical Analysis 2: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; Test type: Superiority; Absolute Risk Difference (%) = 7.5 — The unadjusted absolute risk difference in % between nerinetide and placebo in the no-alteplase subgroup
Statistical Analysis 3: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; Test type: Superiority; Relative Risk Difference (%) = 39.7 — The unadjusted relative risk difference in % between nerinetide and placebo in the no-alteplase subgroup

7. Post Hoc Outcome: Number of Subjects With mRS Score of 0 to 2 in the Alteplase Sub-group
Description: Overall proportion of subjects experiencing a favorable functional outcome 90 days post-randomization, defined as 0 to 2 on the mRS in the sub-group of participants treated with alteplase as part of standard-of-care.
  The modified Rankin Scale (mRS) is a valid and reliable clinician-reported measure of global disability that has been widely applied for evaluating recovery from stroke. It is a scale used to measure functional recovery (the degree of disability or dependence in daily activities) of people who have suffered a stroke. mRS scores range from 0 (best outcome) to 6 (worst outcome), with 0 indicating no residual symptoms; 5 indicating bedbound, requiring constant care; and 6 indicating death.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerinetide, 2.6 mg/kg
Number analyzed (Participants) | 329 | 330
Participants | 216 | 207
Statistical Analysis 1: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.529, Regression, Logistic; Odds Ratio (OR) = 0.887, 95% CI 2-sided [0.612 to 1.286]

8. Post Hoc Outcome: Number of Subjects With NIHSS Score of 0 to 2 in the Alteplase Sub-group
Description: Number of subjects with good neurological outcome, as defined by a score of 0 to 2 on the NIHSS at Day 90 or the last rating in the sub-group of participants treated with alteplase as part of standard-of-care.
  The National Institutes of Health Stroke Scale (NIHSS) is a standardized neurological examination score that is a valid and reliable measure of disability and recovery after acute stroke. Scores range from 0 to 42, with higher scores indicating increasing severity.
Time Frame: 90 days or last rating
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerinetide, 2.6 mg/kg
Number analyzed (Participants) | 329 | 330
Participants | 207 | 191
Statistical Analysis 1: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.181, Regression, Logistic; Odds Ratio (OR) = 0.782, 95% CI 2-sided [0.545 to 1.121]

9. Post Hoc Outcome: Mortality Rate in the Alteplase Sub-group
Description: Mortality rate, as defined by event rate (%) for mortality over the 90-day study period in the sub-group of participants treated with alteplase as part of standard-of-care
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Nerinetide, 2.6 mg/kg
Number analyzed (Participants) | 329 | 330
Participants | 31 | 39
Statistical Analysis 1: Comparison: Placebo vs Nerinetide, 2.6 mg/kg; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.869, Regression, Logistic; Odds Ratio (OR) = 1.050, 95% CI 2-sided [0.588 to 1.874]

ADVERSE EVENTS:
Time Frame: Adverse Events occurring within 30 days of randomization and all Serious Adverse Events up to the end of study visit (Day 90 visit or death) or until the subject was deemed "lost to follow-up" were reported.
Description: All Adverse Events (Serious and Non-Serious) were monitored for the Safety Population, which included all subjects who received any amount of study drug (total of 1101 subjects).
  Adverse Events of Special Interest (AESI) were also collected, and included any Adverse Event which occurred within 2 hours of end of drug infusion and which fall under the standardized MedDRA queries of "Angioedema", "Anaphylactic reaction", "Anaphylactic shock" and terms relating to "hypotension".
Arm/Group | Placebo | Nerinetide, 2.6 mg/kg
All-Cause Mortality (participants affected / at risk) | 74/556 | 64/549
Serious Adverse Events (participants affected / at risk) | 198/554 | 181/547
Other Adverse Events (participants affected / at risk) | 472/554 | 474/547
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=554) | Nerinetide, 2.6 mg/kg (N=547)
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 3
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 6
Atrial flutter (Cardiac disorders) | 1 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 3 | 0
Cardiac arrest (Cardiac disorders) | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 4 | 9
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 2 | 0
Mitral valve stenosis (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 6
Sinus arrest (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Atrial septal defect (Congenital, familial and genetic disorders) | 2 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 1 | 3
Retinal detachment (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 6
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Complication associated with device (General disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 0
Vascular stent occlusion (General disorders) | 2 | 0
Vessel puncture site haematoma (General disorders) | 3 | 1
Vessel puncture site haemorrhage (General disorders) | 0 | 2
Vessel puncture site occlusion (General disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cardiac valve abscess (Infections and infestations) | 0 | 1
Cardiac valve vegetation (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Empyema (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 3 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 6
Pneumonia bacterial (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 6 | 3
Septic shock (Infections and infestations) | 2 | 1
Stoma site abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 5
Urosepsis (Infections and infestations) | 2 | 3
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Cerebral hyperperfusion syndrome (Injury, poisoning and procedural complications) | 0 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Reocclusion (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 5 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 3 | 2
Vascular procedure complication (Injury, poisoning and procedural complications) | 8 | 9
Hepatic enzyme abnormal (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 5 | 4
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 11 | 8
Ischaemic stroke (Nervous system disorders) | 20 | 18
Lacunar stroke (Nervous system disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 4 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Stroke in evolution (Nervous system disorders) | 43 | 36
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 5
Vascular dementia (Nervous system disorders) | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 4 | 0
Mental status changes (Psychiatric disorders) | 1 | 1
Post stroke depression (Psychiatric disorders) | 4 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 3
Azotaemia (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 12 | 19
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1
Loss of personal independence in daily activities (Social circumstances) | 1 | 0
Left atrial appendage occlusion (Surgical and medical procedures) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Brachiocephalic vein thrombosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1
Haematoma (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 7
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 2
Peripheral artery thrombosis (Vascular disorders) | 1 | 2
Peripheral ischaemia (Vascular disorders) | 1 | 1
Varicose vein (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=554) | Nerinetide, 2.6 mg/kg (N=547)
Headache (Nervous system disorders) | 88 | 79
Hemorrhagic Transformation Stroke (Nervous system disorders) | 66 | 60
Hypotension (Vascular disorders) | 54 | 60
Urinary tract infection (Infections and infestations) | 68 | 52
Vascular procedure complication (Injury, poisoning and procedural complications) | 54 | 49
Atrial fibrillation (Cardiac disorders) | 45 | 48
Pyrexia (General disorders) | 47 | 40
Nausea (Gastrointestinal disorders) | 31 | 37
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 28 | 35
Constipation (Gastrointestinal disorders) | 45 | 34
Anemia (Blood and lymphatic system disorders) | 42 | 33
Hypokalaemia (Metabolism and nutrition disorders) | 34 | 33
Vessel puncture site hematoma (General disorders) | 28 | 32
Vomiting (Gastrointestinal disorders) | 36 | 31
Bradycardia (Cardiac disorders) | 32 | 18
Stroke In Evolution (Nervous system disorders) | 54 | 48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT02930018/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT02930018/SAP_001.pdf